CLINICAL TRIAL: NCT05708482
Title: Evaluation of the Effect of Sling and Swing Positions to Pregnant Women in Labour on the Labour Process and Birth Outcomes
Brief Title: Sling and Swing Positions to Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Collaborators: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Nükhet Kaçar, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AnkaraCHBilkent-MH-NK
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Labor; Parturition; Delivery
Keywords: delivery duration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sling-Swing Group (Experimental): 1. While the pregnant woman has 6 cm cervical dilatation examination, the flexible fabric will pass under the arms of the pregnant woman to form a hanger shape. The pregnant woman will be asked to hold the fabric on her feet in a squat and the hanging technique will be applied for 10 minutes. Then, a swing shape will be created in such a way that the flexible fabric will wrap around the chest area of the pregnant woman. The pregnant woman will be asked to hold the fabric in a squat above the knee and the rocking technique will be applied for 10 minutes. Subsequently, uterine contractions, fetal heart rate, fetal head level, position and presence of molding will be evaluated.
  2. Until the completion of the first stage of labor (10 cm cervical dilatation, 100% cervical effacement), this applicant will be experienced by them as the same procedure, hourly.
  3. A Birth Satisfaction Form will be filled at the 2nd hour after delivery..
  Interventions: Other: Sling-Swing Position
- Standard Care Group (No Intervention): 1. While the pregnant woman has 6 cm cervical dilatation examination, uterine contractions, fetal heartbeat, fetal head level, position and presence of molding will be evaluated.
  2. Until the completion of the first stage of labor (10 cm cervical dilatation, 100% cervical effacement), uterine contractions, fetal heartbeat, fetal head level, position and presence of molding will be evaluated every hour.
  3. A Birth Satisfaction Form will be filled at the 2nd hour after delivery. At the end of the study, delivery times and satisfaction of pregnant women will be analyzed.

INTERVENTIONS:
Other: Sling-Swing Position — The device is hammock which look likes a rope
  Arms: Sling-Swing Group

SUMMARY:
It is an experimental and randomized controlled study planned to evaluate the effect of sling-swinging position on the birth experience in vaginal delivery.

DETAILED DESCRIPTION:
In the sample calculation of the study, the sufficient sample size to be studied with a power of 95% based on d=0.8 (large) effect size alpha=0.05 was calculated using the G*Power 3.1.9.4 program, 35 for the application group and 35 for the control group, a total of 70 people.

According to Robson scoring, the midwife can follow the birth process and Pregnant women who are in the active phase of the first stage of labor (5 cm cervical dilatation) are inclusion criterias.

In the study, data have been collected using Introductory Information and Birth Process Follow-up Form and Postpartum Satisfaction Form were developed by the researchers.

For intervention group:

1. While the pregnant woman has 6 cm cervical dilatation examination, the flexible fabric will pass under the arms of the pregnant woman to form a hanger shape. The pregnant woman will be asked to hold the fabric on her feet in a squat and the hanging technique will be applied for 10 minutes. Then, a swing shape will be created in such a way that the flexible fabric will wrap around the chest area of the pregnant woman. The pregnant woman will be asked to hold the fabric in a squat above the knee and the rocking technique will be applied for 10 minutes. The comfort of the pregnant woman will be questioned throughout the procedure. Subsequently, uterine contractions, fetal heart rate, fetal head level, position and presence of molding will be evaluated.
2. Until the completion of the first stage of labor (10 cm cervical dilatation, 100% cervical effacement), the pregnant will be held in the hanging position for 10 minutes and rocking position for 10 minutes, once an hour. Uterine contractions, fetal heartbeat, fetal head level, position and presence of molding will be evaluated after each application, hourly.

For control group:

1. While the pregnant woman has 6 cm cervical dilatation examination, uterine contractions, fetal heartbeat, fetal head level, position and presence of molding will be evaluated.
2. Until the completion of the first stage of labor (10 cm cervical dilatation, 100% cervical effacement), uterine contractions, fetal heartbeat, fetal head level, position and presence of molding will be evaluated every hour.

For Each Group:

A Birth Satisfaction Form will be filled at the 2nd hour after delivery. At the end of the study, delivery times and satisfaction of pregnant women will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* According to Robson scoring, the midwife can follow the birth process.
* Pregnant women who are in the active phase of the first stage of labor

Exclusion Criteria:

* It was decided to deliver by cesarean section due to any indication.
* Pharmacological approach applied
* Any maternal-fetal complication developed
* Those with a height of 150 cm and below
* Pregnant women who want to quit working
* Excluding the inclusion criteria
* Does not know Turkish language (reading-writing-speaking-listening)
* Pregnant women diagnosed with mental and/or auditory disabilities

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Duration of Labor | during labor process
  It is about time as a minute
Satisfaction of Labor | postpartum second hour
  It is about a point which is evaluated by using form. This simple form was developed by researchers. It has five state and its maximum point is 25 and minimum point is 5. The satisfaction increases, the point increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital- Maternity Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is about the ethical process.